CLINICAL TRIAL: NCT00366847
Title: Computer Modeling of Congenital Heart Disease
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 06-149
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Congenital Disorders
Keywords: cardiac; MRI; pediatrics
MeSH Terms: conditions — Congenital, Hereditary, and Neonatal Diseases and Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This proposal is aimed at developing a novel method for modeling and analyzing clinical factors impacting RV function, which can lead to a more reliable, consistent, and comprehensive pre-operative treatment planning. In particular, the proposed work centers on the creation of an accurate and clinically useful heart model with which to quantify, visualize, and interpret several clinical findings that are central to the medical decision-making process. The hypothesis is that by providing clinicians with 3D models that capture numerous relevant patient findings in an integrated, quantitative manner they can make more consistent, reliable, and accurate clinical assessments and may also be able to predict factors complicit in RV dysfunction and impending failure.

DETAILED DESCRIPTION:
The research proposed here is motivated by the need to support pediatric cardiologists in making image-based decisions in the assessment and management of congenital heart disease (CHD). In marked contrast to adult cardiology, which deals almost exclusively with the left ventricle (LV), the function of the RV is associated with a number of life-threatening conditions in pediatrics. These defects include Hypoplastic Left Heart Syndrome (HLHS), Congenitally Corrected Transposition of Great Arteries, Post operative Tetralogy of Fallot, and Double Outlet Right Ventricle.

In particular, a computer model that simulates both the myocardium and blood pool of the right ventricle (RV) is being investigated that can be used to measure clinically useful but diverse parameters of RV blood flow and wall behaviors that previously would require multiple analysis tools to acquire. The model is based on data from MRI studies of patients. Alternate measurement techniques such as ultrasound and catheter pressure measurements are needed to verify the efficacy of the model.

Through a retrospective chart review of CHD patients with defects associated with RV dysfunction, data will be obtained from CHOA over a five year period, June 1, 2001 through May 31, 2006. It will be collected from 10 children aged 0-18 years. Magnetic Resonance images, Ultrasound and catheterization measurements will be collected and analyzed.

Data from MR will be used primarily to determine RV volumetric data. This information will be used to determine RV shape at the different stages of systole and through diastole. The RV shapes are the input to the computer model. The computer model will determine relevant clinical measures such as ejection fraction, pressure measurements, strain rate, and wall thickening based solely on the MR image data. The ultrasound and catheter data will be used as independent sources of verification against the data determined from the computer model. Ultrasound data will be used to compare ejection fraction and wall behavior to the predictive model and catheter data will be used to compare pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

* Choa patients only. Data will be taken from the following patient groups:

  * Normal right ventricular (RV) EF with normal RV size and pulmonary insufficiency (PI)
  * Normal RV EF with dilated RV and PI
  * Reduced RV EF with dilated RV with PI
  * Normal RV EF (pre-operatively) dilated RV and pulmonary valve
  * replacement
  * Reduced RV EF (pre-op) dilated RV and pulmonary valve replacement

Exclusion Criteria:

* Those who do not conform with inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a chart review of patients with heart defects associated with Right Ventricle dysfunction who have received a cardiac MRI at Children's Healthcare of Atlanta between January 1, 1990 and March 14, 2007.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2001-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
RV Function | 1/1/1990- 3/14/2007
  This proposal is aimed at developing a novel method for modeling and analyzing clinical factors impacting RV function, which can lead to a more reliable, consistent, and comprehensive pre-operative treatment planning.

CONTACTS AND LOCATIONS:
Overall Officials: Marijn E Brummer, PhD, Principal Investigator — Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States